CLINICAL TRIAL: NCT03696407
Title: A Non-interventional Retrospective Study to Describe Early Clinical Experience With Cabozantinib in Patients With Advanced Renal Cell Carcinoma in the United Kingdom (UK)
Brief Title: A Non-interventional Retrospective Study to Describe Early Clinical Experience With Cabozantinib in Patients With Advanced Renal Cell Carcinoma (RCC) in the UK
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-GB-60000-017
Record Dates: First submitted 2018-10-03; First posted 2018-10-04 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Advanced Renal Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical experience with cabozantinib is limited in the UK and Ireland and there is anecdotal evidence of there being variability between clinicians in terms of where cabozantinib is used in the treatment pathway. The present study aims to collate and report the experiences of a sample of National Health Service (NHS) Trusts that enrolled patients onto the managed access programme. The study will describe the positioning of cabozantinib in the treatment pathway, associated clinical outcomes and characteristics of patients with advanced RCC receiving cabozantinib in this early clinical experience setting. The results will provide valuable information for collective learning on how to prescribe and manage cabozantinib and its optimal positioning in the patient pathway. Overall, the findings will contribute to a better understanding of how best to manage patients with advanced RCC in routine practice.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of advanced RCC
* Prescribed cabozantinib as part of the Managed Access Programme (MAP) (alive or deceased at study data collection)
* Aged ≥18 years at start of cabozantinib treatment.

Exclusion Criteria:

* Decline or lack the capacity to consent for researcher access to their medical records (if living)
* Hospital medical records are unavailable for review

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Secondary/tertiary care service
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Positioning of cabozantinib in the treatment pathway | 24 months
  Positioning of cabozantinib in the treatment pathway (second line, third line, fourth line or above)
Distribution of cabozantinib starting dose. | Baseline
  Distribution, mean (SD) and median (quartiles) cabozantinib starting dose.
Daily dose during treatment | 24 months
  Mean (SD) and median (quartiles) cabozantinib daily dose during treatment.
Proportion of patients with dose modifications | 24 months
  Proportion of patients with dose modifications and mean (SD) and median (quartiles) number of dose modifications per patient.
Median time to first dose modification | 24 months
Distribution of reasons for dose modifications. | 24 months
Proportion of patients permanently discontinuing cabozantinib. | 24 months
Distribution of reasons for discontinuation of treatment | 24 months
Median duration of cabozantinib treatment (months) | 24 months
Distribution of relevant concomitant treatments | 24 months
  Radiation procedures, denosumab, bisphosphonates.
Distribution of systemic therapies prescribed for advanced RCC after discontinuation of cabozantinib. | 24 months

SECONDARY OUTCOMES:
Distribution of RCC stage and histological type at initial RCC diagnosis | baseline
Time (months) from advanced RCC diagnosis to cabozantinib initiation. | baseline
  Mean (SD) and median (quartiles) time (months
Distribution of RCC stage at cabozantinib initiation. | baseline
Distribution of metastatic sites. | baseline
  Metastatic sites (lung / liver / bone / lymph node / brain / visceral other) documented co-morbidities and distribution of relevant co-morbidities.
Distribution of International Metastatic Renal Cell Carcinoma Database Consortium (IMDC) risk group | baseline
  Distribution of IMDC risk group (favourable, intermediate, poor). From patient's medical records (if documented) or calculated from the individual components (haemoglobin, Karnofsky Performance Status, time from advanced RCC diagnosis to systemic treatment initiation, calcium, neutrophils, platelets).
Progression Free Survival (PFS) | 3, 6, 9, 12, 18 and 24 months and median PFS.
  PFS is defined as the time from cabozantinib initiation until the date of first documented evidence of disease progression or death from any cause. Disease progression is defined as either radiological disease progression (according to RECIST criteria [if documented in routine practice] or other local investigator assessment]) or clinical progression
Overall Survival (OS) | 6, 12, 18 and 24 months
  OS will be measured from both cabozantinib initiation (time from cabozantinib initiation until death from any cause) and from advanced RCC diagnosis (from advanced RCC diagnosis until death from any cause).
Objective Response Rate (ORR) | 3, 6, 9 and 12 months
  ORR defined as the proportion of patients achieving a complete or partial response

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (6):
- United Kingdom (6):
  - Royal Sussex County Hospital, Brighton
  - Addenbrooke's Hospital, Cambridge
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Surrey County Hospital, Guildford
  - St Bartholomew's Hospital, London
  - The Christie Hospital, Manchester